CLINICAL TRIAL: NCT06769243
Title: Cognitive Flexibility and Response to TMS Therapy in Obsessive-Compulsive Disorder
Brief Title: Cognitive Flexibility and Response to TMS Therapy
Acronym: CogFlexTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Beyazit Garip, Director of Gulhane Brain Stimulation Center, Gulhane Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-19
Record Dates: First submitted 2024-12-29; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Obsessive-Compulsive Disorder; Cognitive Flexiblity
Keywords: TMS; Cognitive Felxibility; Obsessive; Compulsive; Treatment Response
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: The treatment-resistant OCD group will be evaluated both before and after TMS treatment. Cognitive flexibility levels of patients will be assessed only prior to the TMS procedure. A control group consisting of healthy participants will be evaluated solely from a neuropsychological and clinical perspective, without undergoing TMS treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Flexibility (Experimental): The TMS protocol was conducted using the MagVenture X100 device. Prior to treatment, a pre-evaluation was performed based on the pre-treatment risk assessment form for patients included in the study. Motor threshold measurement was carried out before the TMS application and repeated weekly. The treatment intensity was set at 100% of the measured motor threshold. As part of the OCD protocol, patients were subjected to 1 Hz rTMS pulses for 300 seconds, with a 60-second intertrain interval, totaling 1200 pulses per session. Each patient received 20 treatment sessions, resulting in a total of 24,000 pulses. The bilateral supplementary motor area (SMA) was targeted. To locate the SMA, after identifying the cranial apex, 15% of the total distance from the front was calculated.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Transcranial Magnetic Stimulation (TMS) is a noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain. It is primarily used to treat OCD, particularly in patients who have not responded well to traditional treatments such as medications or psychotherapy. The most common target is the supplementary motor area (SMA), which has an indirect connection with the Cortico-Striato-Thalamo-Cortical (CSTC) pathway, known to be hyperactive in OCD.
  Another option to target the CSTC pathway is deep TMS, although it is not available in most advanced centers. The magnetic pulses from TMS stimulate or inhibit brain activity in the targeted area, which is believed to help reset or correct neural activity patterns associated with OCD and other psychiatric disorders.
  TMS represents an alternative treatment for those struggling with OCD, offering a non-invasive approach with relatively few side effects and significant potential benefits.

SUMMARY:
Transcranial Magnetic Stimulation (TMS) therapy is an approved and effective treatment option for treatment-resistant obsessive-compulsive disorder. The present study aims to investigate the relationship between cognitive flexibility and TMS treatment. The main question it aims to answer is:

Does cognitive flexibility predict the TMS treatment response rate? Patients will undergo neuropsychological tests to evaluate cognitive flexibility before the TMS application. A clinical scale to assess the severity of obsessive-compulsive symptoms will be administered using psychometric scales both before and after the TMS procedure.

TMS treatment will be applied five days a week for four weeks.

DETAILED DESCRIPTION:
This prospective cohort study aims to investigate the relationship between transcranial magnetic stimulation (TMS) and cognitive flexibility in patients with treatment-resistant obsessive-compulsive disorder (OCD). Treatment-resistant OCD represents a subset of OCD in which patients do not adequately respond to conventional treatments such as cognitive-behavioral therapy (CBT) and selective serotonin reuptake inhibitors (SSRIs). Emerging evidence suggests that TMS, a noninvasive brain stimulation technique, can effectively alleviate symptoms in treatment-resistant OCD. However, its relationship with cognitive flexibility remains poorly understood.

This study seeks to fill this knowledge gap by assessing cognitive flexibility before TMS treatment to identify patients cognitively suitable for this intervention and understand how they respond to TMS. Another important factor to be investigated is whether there are differences between TMS responders and non-responders.

The study will enroll 30 patients diagnosed with treatment-resistant obsessive-compulsive disorder (OCD) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria. Participants will undergo a TMS treatment treatment using the MagVenture™ X100™ device. The treatment protocol will include 20 sessions over four weeks, delivering a total of 24.000 pulses.

The stimulation will target the supplementary motor area (SMA), a region associated with OCD symptom regulation, with parameters optimized to achieve therapeutic effects while minimizing adverse side effects. Motor threshold measurements will be conducted prior to the initiation of treatment and adjusted weekly to ensure consistent treatment intensity.

A control group of 60 healthy participants will undergo a single neuropsychological evaluation for baseline comparison but will not receive TMS treatment or follow-up.

Comprehensive neuropsychological and clinical psychometric assessments will be conducted for all patients prior to the TMS treatment. After completing the 20 sessions of TMS treatment, patients will undergo clinical psychometric evaluations again.

The neuropsychological assessments will include the Wisconsin Card Sorting Test (WCST), Trail Making Test (TMT), and Verbal Fluency (VF) test. Psychiatric assessments will utilize the Yale-Brown Obsessive Compulsive Scale (Y-BOCS), Patient Health Questionnaire (PHQ-9), and Clinical Global Impression-Improvement (CGI-I) scale to evaluate changes in the severity of OCD symptoms.

The primary objective is to determine whether cognitive flexibility in OCD patients plays a role in predicting the response to TMS treatment. Secondary objectives include identifying any differences in cognitive flexibility test results between TMS responders and non-responders.

The primary outcomes will focus on whether cognitive flexibility-defined as the ability to adapt and cope with stress-affects the outcome of TMS treatment. This is particularly important for identifying patients who are likely to benefit from this time-intensive and prolonged treatment. Knowing in advance which patients are unlikely to respond to TMS treatment could help guide them toward alternative therapies, benefiting both patients and physicians.

Additionally, although TMS is highly effective for OCD treatment, literature suggests that up to half of patients do not respond. Understanding whether these non-responders are cognitively inflexible could help identify specific cognitive subtypes of OCD patients. This knowledge would be invaluable for tailoring treatments and improving outcomes for this challenging subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* According to the DSM-5 TR, those diagnosed with Obsessive-Compulsive Disorder (OCD),
* Failure to respond to at least two different antidepressants and anti-obsessive agents at effective doses and durations,
* The condition cannot be better explained by a metabolic or organic disorder,
* No contraindications to treatment were identified based on the risk assessment scale applied before TMS.

Exclusion Criteria:

* Detection of a contraindication for treatment based on the pre-TMS risk assessment form,
* Detection of an epileptic focus in the pre-TMS electroencephalography findings,
* Diagnosis of a psychotic disorder or bipolar mood disorder,
* Active suicidal thoughts and high risk for suicide,
* The participant to be included in the study has a history of alcohol, substance, or stimulant abuse or addiction (excluding cases where they have not used these substances in the last 12 months or have no history of alcohol misuse), based on a semi-structured clinical interview.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
The Effect of Cognitive Flexibility on TMS Treatment Response | From enrollment to the end of treatment at 4 weeks
  The changes in psychometric scales before and after TMS treatment will determine whether a patient is a TMS responder. Cognitive flexibility, measured at the beginning of treatment, may influence the changes in these psychometric scales. This study will examine the relationship between TMS response rate and cognitive flexibility in OCD patients.
Cognitive Flexibility Features in TMS Responders vs. Non-Responders | From enrollment to the end of treatment at 4 weeks
  Cognitive flexibility features in TMS responders will be compared with non-responders and healthy controls. Specific features in responders vs. non-responders will be evaluated in detail. Cognitive flexibility may be identified as a distinguishing factor in OCD subtypes within the non-responder group. This could be useful for navigating treatment options at the beginning of the TMS procedure.
Improvement of the Obsessive-Compulsive Scale: Y-BOCS | From enrollment to the end of treatment at 4 weeks
  A reduction of more than 30% in the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score will be used to evaluate treatment response. The Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) is commonly used to assess the severity of obsessive-compulsive disorder (OCD).The Y-BOCS consists of 10 items, each rated on a scale from 0 (no symptoms) to 4 (extreme symptoms). These items are divided into obsessions (5 items) and compulsions (5 items), allowing for a subscore for each domain (maximum of 20 each). Minimum Score: 0 (indicating no symptoms). Maximum Score: 40 (indicating extreme severity of symptoms)
Changes in PHQ-9 Scores Among Patients with Obsessive-Compulsive Disorder | From enrollment to the end of treatment at 4 weeks
  The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, monitor, and measure the severity of depression. A clinical response is typically defined by a measurable reduction in symptom severity, in depression, a clinical response is defined as a 50% or greater reduction in scores on PHQ-9. The PHQ-9 (Patient Health Questionnaire-9) has the following scoring range: Minimum Score: 0 (indicating no depressive symptoms). Maximum Score: 27 (indicating severe depressive symptoms).
Neuropsychological Test Changes in Obsessive-Compulsive Disorder:WCST | From enrollment to the end of treatment at 4 weeks
  The Wisconsin Card Sorting Test (WCST) is a neuropsychological test designed to evaluate executive functions, including cognitive flexibility, problem-solving, and the ability to adapt to changing rules. It is commonly used in research and clinical settings to assess individuals with neurological or psychiatric conditions
  Measures and Scoring:
  Number of Categories Completed: Indicates how many correct sorting rules the participant identified.
  Perseverative Errors: Reflects the tendency to persist with an incorrect rule despite feedback.
  Non-perseverative Errors: Errors that are not related to the previously learned rule.
  Failure to Maintain Set: Reflects the inability to consistently apply a correct sorting rule.
  Trials to Complete the First Category: Measures the efficiency in initially identifying a rule.
Neuropsychological Test Changes in Obsessive-Compulsive Disorder: TMT A/B | From enrollment to the end of treatment at 4 weeks
  The Trail Making Test (TMT) is a neuropsychological assessment tool used to measure cognitive flexibility, processing speed, and executive functioning.
  TMT-A: Normal Performance: Typically, scores are within 30-60 seconds for healthy adults. Slower Time: Suggests processing speed or attention difficulties, which may be seen in conditions such as ADHD, depression, or neurological impairments.
  TMT-B: Normal Performance: Usually takes 60-150 seconds for healthy adults. Slower Time: A significant delay in TMT-B (compared to TMT-A) can suggest difficulty with task-switching, cognitive flexibility, or executive function, often seen in frontal lobe dysfunction, dementia, Parkinson's disease, or other cognitive impairments.
Memory Performance in Obsessive-Compulsive Disorder: Verbal Fluency Test (VF)" | From enrollment to the end of treatment at 4 weeks
  Verbal Fluency Test (VFT), is a neuropsychological test that measures a person's ability to generate words within a specific category (semantic fluency) or starting with a specific letter (phonemic fluency) in a set amount of time. It is used to assess executive functions, language, and cognitive flexibility.
  Semantic Fluency (Category Fluency): The participant is asked to name as many items as possible within a given category, such as animals or fruits, in 60 seconds.
  Phonemic Fluency (Letter Fluency): The participant is asked to generate as many words as possible that begin with a given letter (e.g., "K", "A", or "S") in 60 seconds.
  Scoring: The score is based on the number of words the participant can generate within the time limit.

SECONDARY OUTCOMES:
Analyzing the Relationship Between Cognitive Flexibility and Symptom Severity | From enrollment to the end of treatment at 4 weeks
  Symptom severity, measured at the beginning of the TMS procedure, may have a relationship with the patient's cognitive flexibility level compared to healthy controls. Symptom severity, assessed using the Yale-Brown Obsessive Compulsive Scale (Y-BOCS), will reflect the clinical severity of OCD symptoms. Understanding any correlation between symptom severity and cognitive flexibility would be beneficial for guiding treatment during the TMS procedure.
Side Effects Assessment | From enrollment to the end of treatment at 4 weeks
  Recording any adverse events or unexpected side effects noted during or after the transcranial magnetic stimulation (TMS) sessions, to evaluate the safety profile of the treatment. There is no standardized method for evaluating the side effects of TMS, a clinician will evaluate the participants for known side effects including changes in hearing, local pain, muscle contractions, headache, non-specific tingling, and discomfort.
Tracking Reduction in Symptom Severity: Yale-Brown Obsessive-Compulsive Scale | From enrollment to the end of treatment at 4 weeks
  Symptom severity in Obsessive-Compulsive Disorder will be evaluated using the Yale-Brown Obsessive Compulsive Scale (Y-BOCS). A 30% reduction in Y-BOCS symptoms will be considered a response to treatment. The Y-BOCS assesses the severity of obsessive-compulsive symptoms, with a minimum score of 0, indicating no obsessive-compulsive symptoms, and a maximum score of 40, indicating extreme severity of obsessive-compulsive symptoms.
Tracking Reduction in Symptom Severity: Patient Health Questionnaire-9 | From enrollment to the end of the treatment at 4 weeks.
  A ≥ 50% reduction in the PHQ-9 score is often considered a clinically significant response to treatment. The PHQ-9 scoring ranges from a minimum score of 0, indicating no depressive symptoms, to a maximum score of 27, indicating severe depressive symptoms. The interpretation of PHQ-9 scores is as follows: 0-4 indicates minimal or no depression, 5-9 indicates mild depression, 10-14 indicates moderate depression, 15-19 indicates moderately severe depression, and 20-27 indicates severe depression.
Drug Side Effect: Common Terminology Criteria for Adverse Events (CTCAE) | From enrollment to the end of treatment at 4 weeks
  The impact of drug side effects on TMS outcomes will be evaluated by assessing the incidence and severity of adverse events using the Common Terminology Criteria for Adverse Events (CTCAE). This standardized tool is commonly used to grade the severity of side effects, ranging from Grade 1 (mild) to Grade 5 (fatal).
  Grade 1: Mild symptoms that do not require intervention. Grade 2: Moderate symptoms that require medical intervention. Grade 3: Severe symptoms that interfere with daily functioning. Grade 4: Life-threatening symptoms requiring urgent medical attention. Grade 5: Death caused by the adverse event.
Drug Side Effect: Visual Analog Scale (VAS) | From enrollment to the end of the treatment at 4 weeks.
  The Visual Analog Scale (VAS) is a commonly used tool for evaluating the intensity of side effects, especially pain, though it can also assess other subjective symptoms such as nausea, fatigue, or dizziness. The VAS consists of a 10 cm long straight line, with one end indicating no symptoms and the other end representing the most severe symptoms possible.
  For assessing pain or side effects, the patient marks a point on the line that reflects the intensity they perceive. The distance from the "no symptoms" end is then measured to determine the severity score.
  0: No pain or side effect 10: Worst possible pain or side effect.

CONTACTS AND LOCATIONS:
Overall Officials: BEYAZIT GARIP, Medical Doctor, Principal Investigator — Gulhane Trainin and Research Hospital
Locations (1):
- Gulhane Training and Research Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IDP) will be shared together with the Clinical Study Report
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be made available immediately after the publication, and will remain available for at least 5 years.
Access Criteria: Anyone who wishes to access the data